CLINICAL TRIAL: NCT04439188
Title: MATCH Treatment Subprotocol P: Phase II Study of PI3K Beta Specific Inhibitor, GSK2636771, in Patients With Tumors With PTEN Loss by IHC
Brief Title: Testing GSK2636771 as a Potential Targeted Treatment in Cancers With PTEN Loss of Expression (MATCH-Subprotocol P)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03143; NCI-2020-03143 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-P (Other: ECOG-ACRIN Cancer Research Group); EAY131-P (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma | interventions — GSK2636771

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (GSK2636771) (Experimental): Patients receive PI3K-beta inhibitor GSK2636771 400 mg PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: PI3K-beta Inhibitor GSK2636771

INTERVENTIONS:
Drug: PI3K-beta Inhibitor GSK2636771 — Given PO
  Other Names: GSK-2636771; GSK2636771

SUMMARY:
This phase II MATCH treatment trial identifies the effects of GSK2636771 in patients whose cancer has a complete loss of PTEN expression. GSK2636771 may block a protein called PI3K-beta, which may be needed for growth of cancer cells with complete loss of PTEN expression. Researchers hope to learn if GSK2636771 will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive PI3K-beta inhibitor GSK2636771 (GSK2636771) 400 mg orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, and then every 6 months for year 3 from study entry.

THE MATCH SCREENING TRIAL:

Please see NCT02465060 for information on the MATCH Screening Protocol and applicable documents.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients must have complete loss of cytoplasmic and nuclear PTEN staining on immunohistochemistry as determined by the MATCH PTEN immunohistochemistry (IHC) assay performed at MD Anderson. Patients can have any PTEN mutation or deletion status, but MUST have PTEN loss by IHC
* Patients must have hemoglobin >= 9 g/dL
* Patients must have a serum creatinine that is < 1.5 x upper limit of normal (ULN) or have a 24-hour creatinine clearance of > 50 mL/min

Exclusion Criteria:

* Patients must not have known hypersensitivity to GSK2636771 or compounds of similar chemical or biologic composition
* Patients must not have tumors harboring co-existing aberrations activating the PI3K/MTOR and MAPK pathways, such as PIK3CA, PIK3R1, BRAF, KRAS and AKT1, TSC1/2, mTOR, NF2, NRAS, HRAS, NF1
* Patients must not have received prior treatment with agents targeting the PI3K beta, AKT, or mTOR:

  * This includes (but is not limited to):

    * mTOR inhibitors: temsirolimus, everolimus, ridaforolimus, sirolimus, salirasib, CC-223, INK128, DS-3078, CC-115, AZD-2014
  * Dual PI3K/mTOR inhibitors: BEZ235, XL-765, GDC 0980, PF-04691502, GSK 2126458, Quinacrine, PKI-587, P-P7170, LY3023414, GDC 0084, DS 7423, CBLC-137

    * Pan-PI3K inhibitors: BKM-120 (buparlisib), PX-866, XL-147, GDC-0941 (pictilisib), BAY-806946, ZSTK-474, WX 037, SRX5000, SRX2523, AMG511, PQR308, BAY 94-9343
    * PI3K inhibitors with beta isoform activity: prior GSK2636771 is not allowed, nor is GS-9820, PQR3XX, KAR4139
  * The following previous treatments are allowed:

    * BYL719 (PI3Kalpha inhibitor)
    * GDC-0032 (PI3Kalpha inhibitor)
    * INK1117 (PI3Kalpha inhibitor)
    * Idelalisib (PI3Kdelta inhibitor)
    * IPI-125 (PI3K gamma delta inhibitor)
    * TGR1202 (PI3Kdelta inhibitor)
    * SRX2558 (PI3Kdelta inhibitor)
    * RP6530 (PI3K gamma delta inhibitor)
    * PWT143 (PI3Kdelta inhibitor)
    * IPI443 (PI3K gamma delta inhibitor)
    * GNE293 (PI3Kdelta inhibitor)
* Patients with a history of interstitial lung disease or pneumonitis are excluded
* Patients must not have any congenital platelet function defects and cannot be on any of the following anti-platelet drugs: clopidogrel, ticlopidine, prasugrel, that act at platelet purinergic receptors

  * Any need for starting anti-platelet therapy in a patient enrolled to this arm will have to be evaluated by the subprotocol chair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Filip Janku, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol P was activated on February 25, 2016. Thirty-five patients were enrolled on EAY131-P between March 21, 2016, and February 17, 2017. All patients were enrolled on the basis of the results from the NCI-MATCH assay.
Pre-assignment Details: Patients who had tumor with complete loss of cytoplasmic and nuclear staining for PTEN with IHC were assigned to sub-protocol P. The mutation status was determined by MATCH central Oncomine assay for all patients in this arm.
Period: Overall Study
Arm/Group | Treatment (GSK2636771)
Started | 35
Started Protocol Therapy | 35
Eligible and Treated (Primary efficacy analysis set) | 32
Completed | 0
Not Completed | 35
Not completed — Ineligible | 3
Not completed — Adverse Event | 4
Not completed — Death | 1
Not completed — Disease Progression | 25
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Patients who were eligible, started protocol therapy were the analyzable patients
Arm/Group | Treatment (GSK2636771)
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 63 [24 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Details about how to define complete response and partial response can be found in the master protocol. 90% two-sided binomial exact confidence interval is calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible and treated
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (GSK2636771)
Number analyzed (Participants) | 32
percentage of participants | 0

2. Secondary Outcome: 6-month Progression-free Survival (PFS) Rate
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS rate is determined
Population: Eligible and treated
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (GSK2636771)
Number analyzed (Participants) | 32
percentage of participants | 3.3 [0.4 to 12.1]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible and treated
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (GSK2636771)
Number analyzed (Participants) | 32
months | 1.8 [1.6 to 2.1]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All patients enrolled were included in the all-cause mortality analysis and in the toxicity analysis.
Arm/Group | Treatment (GSK2636771)
All-Cause Mortality (participants affected / at risk) | 31/35
Serious Adverse Events (participants affected / at risk) | 8/35
Other Adverse Events (participants affected / at risk) | 22/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (GSK2636771) (N=35)
Anemia (Blood and lymphatic system disorders) | 2 (8)
Fatigue (General disorders) | 2 (8)
Diarrhea (Gastrointestinal disorders) | 2 (8)
Nausea (Gastrointestinal disorders) | 1 (8)
Alkaline phosphatase increased (Investigations) | 1 (8)
Dehydration (Metabolism and nutrition disorders) | 1 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (8)
Hypokalemia (Metabolism and nutrition disorders) | 2 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (8)
Insomnia (Psychiatric disorders) | 1 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (8)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (GSK2636771) (N=35)
Anemia (Blood and lymphatic system disorders) | 2 (22)
Fatigue (General disorders) | 8 (22)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (22)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (22)
Bloating (Gastrointestinal disorders) | 2 (22)
Constipation (Gastrointestinal disorders) | 2 (22)
Diarrhea (Gastrointestinal disorders) | 14 (22)
Flatulence (Gastrointestinal disorders) | 2 (22)
Nausea (Gastrointestinal disorders) | 11 (22)
Vomiting (Gastrointestinal disorders) | 6 (22)
Alkaline phosphatase increased (Investigations) | 2 (22)
Creatinine increased (Investigations) | 5 (22)
Lymphocyte count decreased (Investigations) | 2 (22)
Platelet count decreased (Investigations) | 2 (22)
Anorexia (Metabolism and nutrition disorders) | 5 (22)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (22)
Hypokalemia (Metabolism and nutrition disorders) | 2 (22)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (22)
Hyponatremia (Metabolism and nutrition disorders) | 2 (22)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (22)
Dizziness (Nervous system disorders) | 3 (22)
Dysgeusia (Nervous system disorders) | 4 (22)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT04439188/Prot_002.pdf
  • Informed Consent Form (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT04439188/ICF_003.pdf